CLINICAL TRIAL: NCT03024736
Title: Neonatal and Maternal Effects of Buprenorphine and Methadone in the Treatment of Opioid-Maintained Pregnant Women: A Retrospective Cohort Study
Brief Title: Neonatal and Maternal Effects of Buprenorphine and Methadone
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jaye Shyken, MD, Principal Investigator, St. Louis University
Other Study IDs: 26451
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Opioid-maintained Pregnant Women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: buprenorphin — if buprenorphine has better neonatal outcomes compared to methadone in
  the treatment of opioid-maintained pregnant women

SUMMARY:
In this retrospective chart review, the investigators plan to analyze the effects of buprenorphine compared to methadone in opioid-maintained pregnant women. The investigators will evaluate both maternal and neonatal outcomes, with a primary outcome of infant hospital length of stay. The investigators will evaluate patients receiving care in a single setting.

DETAILED DESCRIPTION:
In 2012, 5.4% of pregnant women ages 15 to 44 reported using illicit drugs; however this is lower compared to 11.4% in the non-pregnant population. Illicit drug use is highest in the first trimester (9.0%) and continues to decline as the pregnancy progresses (4.8% 2nd trimester and 2.4% 3rd trimester).

The opioid agents include heroin, codeine, fentanyl, hydrocodone, hydromorphone, meperidine, morphine, methadone, and oxycodone. Patients will experience euphoria during intoxication followed by withdrawal, both of which pose a threat to mother and fetus. During euphoria, there is an increased risk of maternal respiratory depression and fetal growth restriction. During withdrawal, tachycardia, hypertension, nausea, vomiting, and increased metabolic demand can occur, which can cause negative outcomes for the fetus such as spontaneous abortion, preterm labor, premature preterm rupture of membranes, intrauterine growth restriction (IUGR) and intrauterine fetal demise (IUFD). Withdrawing is not ideal in pregnancy due to risks to the baby and high risk of relapse in the mother. Heroin withdrawal can occur within the first 24 hours of birth and usually peaks within 48 to 72 hours, but may take up to 7 days for withdrawal to occur.

At birth, infants born to women using illicit drugs can also go through withdrawal,otherwise known as neonatal abstinence syndrome (NAS). NAS is defined as the hyperactivity of the central and autonomic nervous systems. Clinical presentation depends on duration of opioid use, duration of use prior to delivery, maternal metabolism, and placental metabolism. Symptoms of NAS manifest in the CNS and gastrointestinal (GI) tract. If the mother uses nicotine, stimulants, sedatives, SSRIs, etc, this can also affect withdrawal, as all of these agents cause fetal withdrawal as well. Clinicians in the United States primarily use the modified Finnegan's Neonatal Abstinence scoring tool to assess for signs and symptoms and severity of NAS. This tool evaluates 21 items in the areas of CNS disturbances, GI disturbances, and metabolic/vasomotor/respiratory disturbances. Scores can range from 0 to 44 with a score > 8 indicating need of pharmacologic treatment.5 Medication treatment is used to relieve moderate to severe signs of NAS and to prevent complications and may include an opioid, barbiturate, benzodiazepine, clonidine, or chlorpromazine. Methadone has been the standard of treatment for opioid addiction during pregnancy since the 1970s. Methadone is a full mu-agonist that can be used for analgesia or maintenance of opioid addiction. Methadone is dispensed on a daily basis by a registered substance abuse treatment program and is usually started at 10 to 30 mg/day. Methadone can cause serious adverse events such as respiratory depression, QTc prolongation, hypotension, and sedation, with other adverse events including lightheadedness, dizziness, nausea, vomiting, and diaphoresis. Infants exposed to methadone usually experience withdrawal within the first 72 hours, but can occur within the first two weeks and can last for several days to weeks. Recently there has been increasing evidence for the use of buprenorphine in pregnancy due to the potential of less neonatal abstinence syndrome (NAS). Buprenorphine is a partial mu agonist that is indicated for the treatment of opioid dependence with typical doses of 2 to 24 mg. Infants exposed to buprenorphine usually experience withdrawal within 12 to 48 hours, peaks between 72 and 96 hours, and resolves by 7 days.2 Like methadone, there are still risks of respiratory depression, central nervous system (CNS) depression, and hypotension. There is a lower risk of overdose, fewer drug interactions, and does not need to be dispensed daily at clinic, making it a more favorable option over methadone. Buprenorphine does require additional registration for providers to prescribe it, but can be filled at any pharmacy.

The PROMISE trial is a randomized, double-blind, double-dummy, parallel-group controlled trial that was designed to compare methadone and buprenorphine for the treatment of opioid-dependent pregnant patients. A total of 30 patients were enrolled who received methadone or buprenorphine with dosing based on compliance, urine samples, and patient report of withdrawal symptoms and cravings.

The primary outcomes analyzed were number of neonates requiring morphine for NAS, peak NAS score, total amount of morphine given, and total days of neonatal hospital stay. There were several secondary neonatal and maternal outcomes as well. Neonatal length of stay was the only statistically significant outcome, with a difference of 1.3 days in favor of buprenorphine (p= 0.021). There was no difference in adverse events amongst the two groups. This trial was limited due to its small size, but supported the need for a larger trial.8

The MOTHER trial is a multi-center, randomized, double-blind, double-dummy trial that was designed to compare methadone and buprenorphine for the treatment of opioid-dependent pregnant patients. A total of 175 patients were enrolled and received methadone or buprenorphine with dosing based on compliance, urine samples, and patient report of withdrawal symptoms and cravings.

The primary outcomes analyzed were number of neonates requiring treatment for NAS, peak NAS score, total amount of morphine needed for treatment of NAS, length of neonatal hospital stay, and head circumference. There were several secondary neonatal and maternal outcomes measured as well. The total amount of morphine needed and neonatal length of stay were statistically significant. Neonates taking buprenorphine required 1.1 ± 0.7 mg morphine, whereas the methadone group required 10.4 ±2.6 mg morphine (p = 0.0091). The buprenorphine group had a shorter length of stay of 10.0 ± 1.2 days compared to 17.5 ± 1.5 days in the methadone group (p = 0.0091). In regards to secondary outcomes, duration of treatment was significant favoring buprenorphine (4.1 vs. 9.9 days, p = 0.003125). None of the secondary maternal outcomes were statistically significant. The methadone group had a higher incidence of non-serious maternal events and non-serious cardiovascular events. This trial supports that buprenorphine is a safe and effective treatment for opioid dependence in pregnant women.

Based on the aforementioned studies, the investigators established a clinic which has been prescribing buprenorphine for the treatment of opioid dependence for a small group of patients. Patients who are opioid-dependent were evaluated to see if buprenorphine is the best option for them. There is also a prescribing regulation in the first year that limits the provider to prescribing buprenorphine to 30 patients. The remainder of patients has been treated with methadone.

The clinic is multi-disciplinary, and the patients are seen by the maternal fetal medicine specialist, a nurse practitioner, a pharmacist, the social services department, a nurse coordinator, a neonatologist, a lactation nurse, the anesthesia department, and a dietician throughout the pregnancy. Patients enrolled in the clinic must receive all of their obstetric care through the clinic and should deliver within the same health system. Patients starting buprenorphine are initiated in clinic if they are in the first or second trimesters, but admitted for monitoring during buprenorphine induction if 24 weeks or further. After buprenorphine induction, patients are seen weekly for 4 weeks, then every other week over 6 weeks, then every 4 weeks thereafter and as needed for traditional prenatal care needs. Patients must also attend counseling and narcotics anonymous meetings. Once the patient delivers, they are seen twice in the 6 weeks post-partum.

In this retrospective chart review, the investigators plan to analyze the effects of buprenorphine compared to methadone in opioid-maintained pregnant women. The investigators will evaluate both maternal and neonatal outcomes, with a primary outcome of infant hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* patients on buprenorphine or methadone.
* pregnant

Exclusion Criteria:

* Not meeting inclusion criteria

Ages: 13 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Gender: Female ethnic background: all age 13-55yrs of age
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
infant hospital length of stay | 1 year
  The investigators will evaluate both maternal and neonatal outcomes, with a primary outcome of infant hospital length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Jaye Shyken, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No